CLINICAL TRIAL: NCT04986696
Title: A Phase I, First-in-human, Dose Finding Study of High Dose Rate Radiotherapy in Patients With Skin Metastases From Melanoma
Brief Title: Irradiation of Melanoma in a Pulse
Acronym: IMPulse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Jean Bourhis, Prof., MD, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0023-IMPulse-2020
Record Dates: First submitted 2021-07-02; First posted 2021-08-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Metastasis From Malignant Melanoma of Skin (Diagnosis)
Keywords: FLASH therapy; melanoma
MeSH Terms: conditions — Disease; Melanoma

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation of FLASH therapy in skin metastases of small volume (≤ 30 cc) (Experimental): 7 dose levels (22 Gy; 24 Gy; 26 Gy; 28 Gy, 30 Gy, 32 Gy and 34 Gy)
  Interventions: Device: FLASH therapy
- Dose escalation of FLASH therapy in skin metastases of large volume (> 30 and ≤ 100 cc) (Experimental): 7 dose levels (22 Gy; 24 Gy; 26 Gy; 28 Gy, 30 Gy, 32 Gy and 34 Gy)
  Interventions: Device: FLASH therapy

INTERVENTIONS:
Device: FLASH therapy — Dose escalation of high dose rate radiotherapy (FLASH therapy) as single dose treatment for skin melanoma metastases that progress locally despite systemic treatments.
  Other Names: high dose rate radiotherapy

SUMMARY:
This is a single center phase I, first-in-human, dose escalation study of FLASH therapy in patients with metastases of melanoma.

The trial is based on escalating single doses of FLASH therapy administered to skin melanoma metastases using the Mobetron® with high dose rate (HDR) functionality.

The aim of the study is to evaluate a dose escalation of high dose rate radiotherapy (FLASH therapy) as single dose treatment for skin melanoma metastases that progress locally despite systemic treatments. Melanoma is a typically radio-resistant tumor type, which can justify such a dose escalation with a new type of radiotherapy that appears much better tolerated than conventional radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed study Informed Consent Form
2. Karnofsky Performance Status (KPS) ≥ 50
3. Age ≥ 18 years
4. Patients with metastatic melanoma and multiple skin metastases with a documented clinical progression despite the systemic treatments (chemotherapy, and/or Programmed cell death 1 (PD1), cytotoxic T-lymphocyte antigen-4 (CTLA4) inhibitors or tyrosine kinase inhibitors (TKIs), such as v-raf murine sarcoma viral oncogene homolog B1 (BRAF) or mitogen-activated extracellular signal-regulated kinase (MEK) inhibitors)
5. The size of the treated lesions should be ≤ 5.5 cm in diameter and ≤ 2.8 cm thick (caliper-based measurement)
6. The treated lesions should be at least 5 cm apart and must not be located on the face.
7. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (urine or serum) during screening
8. WOCBP must use a contraceptive method

Exclusion Criteria:

1. Previous radiotherapy in the treated area
2. Concomitant auto-immune disease with skin lesions
3. Concomitant use of radio-sensitizer drug
4. Women who are pregnant
5. Current, recent (within 10 days prior start of study treatment), or planned participation in an experimental drug study. During the 4 weeks DLT period, the patient will not be able to participate to any other clinical study.
6. Any serious underlying medical condition that could interfere with study treatment and potential adverse events
7. Any mental or other impairment that may compromise compliance with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) or recommended phase II dose (RP2D), separately for skin metastases of small and large volumes. | from Day 1 to Day 28
  Acute safety (dose limiting toxicity, DLT) of the high dose rate radiotherapy (RT) procedure (for each dose level) will be evaluated during the 4 weeks post-treatment using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0).

SECONDARY OUTCOMES:
Percentage of patients with Hemorrhage related to the treated lesions, assessed visually by the investigator | At each visit, from screening to 12 months post-treatment
  Hemorrhage will be visually assessed (presence/abscence)
Percentage of patients with Skin ulceration related to the treated lesions, assessed visually by the investigator | At each visit, from screening to 12 months post-treatment
  Skin ulceration will be visually assessed (presence/abscence)
Percentage of patients with Pain related to the treated lesions, assessed with analogic visual pain scale | At each visit, from screening to 12 months post-treatment
  Pain will be assessed using an analogic visual pain scale (score from 1 to 10)
Local response of metastases "in the radiation field", measured with calipers | At screening, Day 1, at weeks 1, 3, 4, and 6 post-treatment; at months 3, 6, and 12 post-treatment; and at local progression
  Irradiated lesions will be measured with calipers. Local response of metastases in the radiation field will be calculated as rate over all treated lesions and will be compared between small versus large volume lesions within each dose level.
Frequency of Late side effects observed "in radiation field" | ≥ 6 months post-treatment
Blinded Imaging Central Review (BICR) of photographs evaluating both tumor response and "in radiation field" normal tissue responses around the treated tumors | From Day 1 up to 12 months post-treatment
  A baseline photograph will be taken the day of the treatment in a pre-therapeutic setting with skin delineation of the lesion. Then photos will be repeated at 1 (+/-2d), 3 (+/-2d), 4 (+/-3d), 6 (+/-3d) weeks after treatment, then at 3 (+/-7d), 6 (+/-14d), 12 (+/-14d) months and at progression.
Optical coherence tomography (OCT) examination of the irradiated skin compared to the normal non-irradiated skin | at 4 weeks, 6 months and 12 months post-treatment
  Epidermis thickness and roughness; plexus depth; number and size of vessels; number and size of hairs, will be compared between irradiated skin and normal non-irradiated skin
Frequency of late adverse events (within 12 months post-treatment) for each dose | within 12 months post-treatment
  Long-term safety of RT procedure will be measured as recording of late adverse events (CTCAE v5.0)

OTHER OUTCOMES:
Observation of a potential Abscopal Effect with evidence of tumor regression on metastases outside of the radiation field, measured with a caliper for cutaneous lesion or on radiological images for other lesions | within 12 months post-treatment (at 1, 3, 4, 6 weeks post-treatment; at 3, 6, 12 months post-treatment; at progression)
  Observation of a potential Abscopal Effect with evidence of tumor regression on metastases outside of the radiation field, measured with a caliper for cutaneous lesion or on radiological images for other lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourhis, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Maity A, Koumenis C. Shining a FLASHlight on Ultrahigh Dose-Rate Radiation and Possible Late Toxicity. Clin Cancer Res. 2022 Sep 1;28(17):3636-3638. doi: 10.1158/1078-0432.CCR-22-1255. PMID 35736814